CLINICAL TRIAL: NCT07374939
Title: Medical Cannabis for Nausea in Patients Receiving Moderately or Highly Emetogenic Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Luke Peppone, Associate Professor - Department of Surgery, Cancer Control (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00011238
Record Dates: First submitted 2026-01-16; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Nausea and Vomiting Chemotherapy-Induced
Keywords: medical cannabis; chemotherapy-induced nausea and vomiting; nausea; nausea and vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Medical Marijuana

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate use (Experimental): Participants randomized to the Immediate Use arm will receive New York State medical cannabis certification and initiate medical cannabis use during their first on-study chemotherapy cycle, in addition to standard guideline-recommended antiemetic therapy. Participants will use medical cannabis primarily during the four days surrounding chemotherapy administration, corresponding to the acute and delayed nausea period. Cannabis will be administered by vaporization using a standardized device, dose limits, and schedule. Participants will complete daily nausea and vomiting diaries, cannabis use logs, and symptom questionnaires, and will provide blood samples once per chemotherapy cycle. Outcomes in this arm will be compared to the delayed-use arm to evaluate the preliminary efficacy, safety, and feasibility of medical cannabis for chemotherapy-related nausea.
  Interventions: Drug: Medical Cannabis
- Delayed use (Active Comparator): Participants randomized to the Delayed Use arm will receive standard guideline-recommended antiemetic therapy alone during their first on-study chemotherapy cycle and will not use medical cannabis during this initial evaluation period. This cycle will serve as the comparison condition for nausea outcomes. After completion of the first cycle assessments, participants will receive New York State medical cannabis certification and will initiate medical cannabis use during the subsequent chemotherapy cycle. Cannabis will be administered by vaporization using a standardized device, dose limits, and schedule, primarily during the four days surrounding chemotherapy administration. Participants will complete daily nausea and vomiting diaries, cannabis use logs, symptom questionnaires, and provide blood samples once per chemotherapy cycle to evaluate changes after cannabis initiation.
  Interventions: Drug: Medical Cannabis

INTERVENTIONS:
Drug: Medical Cannabis — Medical cannabis will be used as an adjunct to standard guideline-recommended antiemetic therapy for chemotherapy-related nausea. Participants will obtain state-certified medical cannabis products through a New York State-licensed dispensary and self-administer cannabis via vaporization using a standardized device. Dose limits and timing of use will be guided by the study protocol to promote consistency while allowing individualized use. Medical cannabis will be used during the acute and delayed nausea period, defined as Days 1 through 4 following chemotherapy administration. Participants randomized to the Immediate Use arm will initiate cannabis use during their first on-study chemotherapy cycle, whereas participants randomized to the Delayed Use arm will initiate cannabis use after completion of the first cycle. Cannabis use patterns, nausea and vomiting symptoms, adverse effects, and patient-reported outcomes will be recorded using participant-completed diaries and questionnaires.

SUMMARY:
Many people receiving chemotherapy experience nausea despite standard anti-nausea medications. Medical cannabis is commonly used to help manage nausea, but there is limited scientific evidence about its effectiveness when used alongside modern chemotherapy treatments.

This study will evaluate whether medical cannabis can reduce nausea in adults receiving moderately or highly nausea-causing chemotherapy. Participants will be randomly assigned to start medical cannabis either immediately or after one chemotherapy cycle, allowing comparison of symptoms with and without cannabis use. All participants will continue their usual anti-nausea medications.

The study will also examine effects on vomiting, appetite, pain, fatigue, sleep, mood, quality of life, and inflammation. Results from this pilot study will help determine the safety, feasibility, and potential benefits of medical cannabis for chemotherapy-related nausea and guide future larger clinical trials.

DETAILED DESCRIPTION:
Many people receiving chemotherapy experience nausea, even when they are given standard anti-nausea medications. Vomiting is now often well controlled, but nausea, especially nausea that occurs one or more days after chemotherapy, remains a major problem. Nausea can interfere with daily activities, reduce appetite, worsen quality of life, and sometimes lead to dehydration or delays in cancer treatment. New approaches are needed to better manage chemotherapy-related nausea.

Medical cannabis is commonly used by patients to help with nausea, appetite, sleep, pain, and other treatment-related symptoms. Although cannabis is legal for medical use in many U.S. states and cancer is a qualifying condition, there is limited scientific evidence about how well cannabis works for chemotherapy-related nausea when used alongside modern anti-nausea medications. More research is needed to understand its benefits, risks, and how it may best be used.

The purpose of this study is to collect early (pilot) data on whether medical cannabis can reduce nausea in adults receiving moderately or highly nausea-causing chemotherapy. The study will also examine whether cannabis affects vomiting, appetite, fatigue, sleep, pain, nerve pain, mood, and quality of life. In addition, blood samples will be collected to explore whether cannabis is associated with changes in inflammation related to cancer treatment.

About 50 adults with cancer who are receiving chemotherapy will take part in this study at the University of Rochester Medical Center. Participants must be 21 years of age or older, experiencing significant nausea despite standard anti-nausea medications, and receiving chemotherapy that commonly causes nausea. People with certain medical or psychiatric conditions, recent cannabis use, or lung disease will not be eligible for safety reasons.

Participants will be randomly assigned to one of two groups. One group will begin using medical cannabis during their first study chemotherapy cycle, while the other group will continue usual care for one cycle and then begin using medical cannabis during the next cycle. This delayed-start approach allows each participant to be compared to their own experience before and after cannabis use. All participants will continue to receive their prescribed anti-nausea medications throughout the study.

Medical cannabis will be obtained through a state-licensed dispensary and used primarily during the four days surrounding each chemotherapy treatment, when nausea is most likely to occur. Cannabis will be used with a standardized vaporization device to help ensure consistent dosing. Participants will keep daily diaries to record nausea, vomiting, cannabis use, and any side effects. They will also complete questionnaires about symptoms, mood, and quality of life. Blood samples will be collected once per chemotherapy cycle during routine lab visits.

Possible risks include side effects of cannabis such as dizziness, anxiety, sleepiness, or difficulty concentrating, as well as minor risks from blood draws such as bruising or lightheadedness. Participants will be given safety instructions, including avoiding driving after cannabis use. There may or may not be direct benefit to participants, but the information gained may help improve nausea management for future cancer patients.

This study will provide important early evidence about the safety, feasibility, and potential benefits of medical cannabis for chemotherapy-related nausea and related symptoms, and will help guide larger future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cancer with no previous chemotherapy treatments (aside from current treatment)
* Be scheduled to receive treatment with a chemotherapeutic agent that is classified by the National Comprehensive Cancer Network (NCCN) as having a high emetogenic potential (>90% incidence) or moderate emetogenic potential (30-90% incidence).
* Must be scheduled for a minimum of 3 additional chemotherapy cycles at the time of enrollment.
* Chemotherapy agents may be given intravenously or orally.
* Chemotherapy cycles must be at least two weeks apart.
* For the purposes of this study, Day 1 is defined as the day of chemotherapy administration.
* Chemotherapy may be for adjuvant, neoadjuvant, curative, or palliative intent.
* Highly emetogenic - common types of chemotherapy

  * AC combination defined as any chemotherapy regimen that contains an anthracycline and cyclophosphamide
  * Carboplatin AUC ≥4
  * Carmustine >250 mg/m2
  * Cisplatin
  * Cyclophosphamide >1,500 mg/m2
  * Dacarbazine
  * Doxorubicin ≥60 mg/m2
  * Epirubicin >90 mg/m2
  * Ifosfamide ≥2 g/m2 per dose
  * Mechlorethamine
  * Streptozocin
* Moderately emetogenic - common types of chemotherapy:

  * Aldesleukin >12-15 million IU/m2
  * Amifostine >300 mg/m2
  * Arsenic trioxide
  * Azacitidine
  * Bendamustine
  * Busulfan
  * Carboplatin AUC <4
  * Carmustined ≤250 mg/m2
  * Clofarabine
  * Cyclophosphamide ≤1500 mg/m2
  * Cytarabine >200 mg/m2
  * Dactinomycin
  * Daunorubicin
  * Dual-drug liposomal encapsulation of cytarabine and daunorubicin
  * Dinutuximab
  * Doxorubicind <60 mg/m2
  * Epirubicind ≤90 mg/m2
  * Idarubicin
  * Ifosfamided <2 g/m2 per dose
  * Interferon alfa ≥10 million IU/m2
  * Irinotecan
  * Irinotecan (liposomal)
  * Melphalan
  * Methotrexated ≥250 mg/m2
  * Oxaliplatin
  * Temozolomide
  * Trabectedin
* Be willing to commit to the suggested medication dosing and delivery method, completing evaluation instruments, and attending all study visits.
* Be able to understand English (all assessment instruments are in English).
* Be 21 years of age or older.
* Give informed consent.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, or abstinence) for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.

Exclusion Criteria:

* Participants must not:
* Use of any THC-containing cannabis products within 30 days prior to enrollment, verified by participant self-report.

Allowable: Use of hemp-derived CBD products containing < 0.3 % THC is permitted, consistent with the 2018 Agriculture Improvement Act (federal definition of hemp). Use of CBD products will be documented in baseline case report forms.

* Have any allergies to cannabis or contraindication for cannabis.
* Have an active or recent (< 6 months) substance use disorder, as determined by medical history.
* Have recently quit smoking (< 6 months) or are actively engaged in a smoking-cessation program.
* Have a history of severe anxiety or paranoia on prior exposure to cannabis.
* Have a previous diagnosis of bipolar disorder or schizophrenia.
* Be pregnant or nursing.
* Have had a prior stroke.
* Have moderate or severe chronic obstructive pulmonary disease (COPD), defined as FEV₁ < 50 % predicted or current use of home supplemental oxygen.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Average and Maximum Nausea Severity as Measured by the Nausea and Vomiting Diary | Days 1-4 following chemotherapy administration during up to 3 on-study chemotherapy cycles (Day 1 defined as the day of chemotherapy administration; each chemotherapy cycle is 14-28 days, depending on regimen)
  Average nausea severity will be measured using a participant completed nausea and vomiting diary. Nausea severity is rated on an 11 point numeric scale anchored by "Not at all nauseated" (0) and "Extremely nauseated" (10). Average nausea is calculated as the mean of up to 15 assessment points, including afternoon, evening, and night on Day 1 and morning, afternoon, evening, and night on Days 2 through 4. Higher scores indicate greater nausea severity. Scores will be set to missing if 11 or more of the 15 assessments are missing.
  Maximum nausea severity will be measured using a participant-completed nausea and vomiting diary. Nausea severity is rated on an 11-point numeric scale anchored by "Not at all nauseated" (0) and "Extremely nauseated" (10). Maximum nausea is defined as the highest nausea rating reported across the same 15 assessment points.
Number of Emesis Episodes Recorded in the Nausea and Vomiting Diary | Days 1-4 following chemotherapy administration during up to 3 on-study chemotherapy cycles (Day 1 defined as the day of chemotherapy administration; each chemotherapy cycle is 14-28 days, depending on regimen)
  Emesis episodes will be recorded daily by participants using the nausea and vomiting diary. The outcome is the total number of vomiting episodes recorded during the assessment period.

SECONDARY OUTCOMES:
Complete Protection From Chemotherapy Induced Nausea and Vomiting | Days 1-4 following chemotherapy administration during up to 3 on-study chemotherapy cycles (Day 1 defined as the day of chemotherapy administration; each chemotherapy cycle is 14-28 days, depending on regimen)
  Complete protection is defined as no emesis, no use of additional rescue therapy, and no significant nausea defined as a nausea score of 2 or less on a 0 to 10 numeric rating scale. The outcome will be reported as the proportion of participants meeting these criteria.
Complete Control of Chemotherapy Induced Nausea and Vomiting | Days 1-4 following chemotherapy administration during up to 3 on-study chemotherapy cycles (Day 1 defined as the day of chemotherapy administration; each chemotherapy cycle is 14-28 days, depending on regimen)
  Complete control is defined as no emesis, no use of additional rescue therapy, and no nausea defined as a nausea score of 0 on a 0 to 10 numeric rating scale.
Complete Response to Chemotherapy Induced Nausea and Vomiting | Days 1-4 following chemotherapy administration during up to 3 on-study chemotherapy cycles (Day 1 defined as the day of chemotherapy administration; each chemotherapy cycle is 14-28 days, depending on regimen)
  Complete response is defined as no emesis and no use of additional rescue therapy. The outcome will be reported as the proportion of participants meeting these criteria.
Change in Appetite as Measured by the University of Rochester Cancer Center (URCC) Symptom Inventory | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Appetite will be assessed using the URCC Symptom Inventory. Appetite is measured on an 11 point numeric scale anchored by "Not at all hungry" (0) and "Extremely hungry" (10). Higher scores indicate greater appetite.
Change in Appetite Related Quality of Life as Measured by the Functional Assessment of Anorexia Cachexia Therapy Questionnaire | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Appetite related quality of life will be measured using the Functional Assessment of Anorexia Cachexia Therapy questionnaire, a validated instrument designed to assess quality of life and anorexia or cachexia related concerns. Higher scores indicate better appetite related quality of life.
Change in Anxiety Severity as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Anxiety severity will be measured using the PROMIS Anxiety Short Form. PROMIS T scores are standardized to a mean of 50 and a standard deviation of 10, with higher scores indicating greater anxiety severity.
Change in Depressive Symptoms as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Depressive symptoms will be measured using the PROMIS Depression Short Form. PROMIS T scores are standardized to a mean of 50 and a standard deviation of 10, with higher scores indicating greater depressive symptom severity.
Change in Fatigue as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Fatigue severity will be measured using the PROMIS Fatigue Short Form. PROMIS T scores are standardized to a mean of 50 and a standard deviation of 10, with higher scores indicating greater fatigue severity.
Change in Pain Interference as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Pain interference will be measured using the PROMIS Pain Interference Short Form. PROMIS T scores are standardized to a mean of 50 and a standard deviation of 10, with higher scores indicating greater pain interference.
Change in Physical Function as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Physical function will be measured using the PROMIS Physical Function Short Form. PROMIS T scores are standardized to a mean of 50 and a standard deviation of 10, with higher scores indicating better physical function.
Change in Sleep Disturbance as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Sleep disturbance will be measured using the PROMIS Sleep Disturbance Short Form. PROMIS T scores are standardized to a mean of 50 and a standard deviation of 10, with higher scores indicating greater sleep disturbance.
Change in Ability to Participate in Social Roles and Activities as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Ability to participate in social roles and activities will be measured using the PROMIS Ability to Participate in Social Roles and Activities Short Form. PROMIS T scores are standardized to a mean of 50 and a standard deviation of 10, with higher scores indicating better social participation.
Change in Pain Intensity as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Item | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Pain intensity will be measured using a single PROMIS pain intensity item rated on a numeric scale ranging from 0 no pain to 10 worst imaginable pain. Higher scores indicate greater pain intensity.
Change in Cognitive Function as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function Short Form | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Perceived cognitive function will be measured using the PROMIS Cognitive Function Short Form. PROMIS T scores are standardized with higher scores indicating better cognitive function.
Change in Concerns About Death and Dying as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Health-Related Quality of Life in Neurological Disorders (HDQLIFE) Concern With Death and Dying Scale | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Concerns related to death and dying will be measured using the PROMIS HDQLIFE Concern With Death and Dying Short Form. Higher scores indicate greater concern.
Change in Health Related Quality of Life as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Preference Summary Score | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Health related quality of life will be measured using the PROMIS Preference summary score, a preference based utility score derived from multiple PROMIS domains and calculated using the MultiAttribute Utility Theory method. Higher scores indicate better health related quality of life.
Change in Peripheral Neuropathic Pain as Measured by the EORTC CIPN 20 Questionnaire | Baseline (within 7 days before chemotherapy) and Day 4 following chemotherapy during Cycles 1 and 3; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Peripheral neuropathic pain will be measured using the European Organisation for Research and Treatment of Cancer Chemotherapy Induced Peripheral Neuropathy 20 item questionnaire. Higher scores indicate greater neuropathic symptom severity.
Change in Psychological Distress as Measured by the NCCN Distress Thermometer | Baseline (within 7 days before chemotherapy) to Day 4 after chemotherapy during up to 3 cycles; post-cycle questionnaires completed on Day 4 or within 48 hours (Day 1 = chemotherapy; cycles 14-28 days).
  Psychological distress will be measured using the National Comprehensive Cancer Network Distress Thermometer, an 11 point scale ranging from 0 no distress to 10 extreme distress. Higher scores indicate greater distress.
Subjective Drug Effects as Measured by the Drug Effects Questionnaire | Day 4 following chemotherapy during Cycle 3 only; questionnaire completed on Day 4 or within 48 hours thereafter (Day 1 defined as the day of chemotherapy administration; cycles are 14-28 days).
  Subjective drug effects will be measured using the Drug Effects Questionnaire, which assesses perceived strength of substance effects and desirability of substance effects using numeric rating scales. Higher scores indicate stronger or more desirable subjective effects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome analyses will be made available upon reasonable request. Shared data will include analyzable datasets necessary to reproduce reported results.